CLINICAL TRIAL: NCT05520606
Title: Minimally Invasive Versus Open for Pancreatoduodenectomy：an Retrospective, Observational, Multicenter Real-world Study
Brief Title: Laparoscopic Pancreatoduodenectomy Versus Open Pancreatoduodenectomy
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Professor in Surgery, Chief Physician, Director of Surgical Supervision Department, Deputy Director of Institute of Hepatobiliary&Pancreatic, Director of Department of Biliary-Pancreatic Surgery, Tongji Hospital
Other Study IDs: TJDBPS11
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Resectable Lesions Located in the Pancreatic Head or Periampullary Region
Keywords: laparoscopic; minimally invasive; open resection; Pancreatoduodenectomy
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- minimally invasive surgery: laparoscopic pancreatoduodenectomy.
  Interventions: Procedure: pancreatoduodenectomy
- open surgery: open pancreatoduodenectomy
  Interventions: Procedure: pancreatoduodenectomy

INTERVENTIONS:
Procedure: pancreatoduodenectomy — Pancreatoduodenectomy (Whipple surgery) is a complex surgical procedure and has been accepted as the gold standard treatment for resectable lesions of the pancreatic head and periampullary region

SUMMARY:
This is a single, retrospective, real-world study to investigate the surgical outcomes of minimally invasive pancreatoduodenectomy and open pancreatoduodenectomy, with the perioperative characteristics and long-term overall survival being compared. The investigators aimed to find out whether the minimally invasive surgery is safe and feasible for resectable lesions located in the pancreatic head and periampullary region. And the investigators also want to find out patients with what kind of characteristic can be benefit from the minimally invasive surgery compared with the open approach.

DETAILED DESCRIPTION:
Pancreatoduodenectomy (Whipple surgery) is a complex surgical procedure and has been accepted as the gold standard treatment for resectable lesions of the pancreatic head and periampullary region.To date, how surgeons can safely pass the learning curve of laparoscopic pancreatoduodenectomy (LPD) without potentially harming patients remains a question. Around this topic, the investigators designed real-world study in a single center to retrospectively collect the PD surgeries since July 2014. The investigators aimed to find out whether the minimally invasive surgery is safe and feasible for resectable lesions located in the pancreatic head and periampullary region. And the investigators also want to find out patients with what kind of characteristic can be benefit from the minimally invasive surgery compared with the open approach. Besides, the investigators also want to investigate the clinical characteristics of patients and perioperative outcomes of LPD procedures and aimed to develop and validate a difficulty scoring system for patient selection which could help facilitate a comprehensive and security understanding of LPD for surgeon during different stage of the learning curve.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years.
2. Patients underwent PD surgeries.

Exclusion Criteria:

1. Peritoneal seeding or metastasis to distant sites;
2. Incomplete clinical data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent PD surgeries in Tongji Hospital since January 2014 .
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Postoperative length of stay | up to 90 days
  defined as the time from being admitted to hospital to discharge

SECONDARY OUTCOMES:
Overall survival | through study completion, an average of 5 year
  defined as the duration from the first day after surgery to either the date of death or the last follow-up
Operation time | intraoperative
  defined as the time from skin incision or trocar placement to complete skin closure
postoperative complications | up to 90 days
  Postoperative complications were reviewed within 90 days after surgery and graded according to Clavien-Dindo (CD) classification system. Postoperative biliary leakage, hemorrhage, and liver failure. Wound infection was defined as purulent drainage from the incision or/and positive findings of culture of the fluid or tissue aseptically obtained from the incision.
Reoperation within 90 days | up to 90 days
  defined as any reoperation within 90 days
Mortality | up to 90 days
  defined as any death within 30 days and 90 days, respectively
Readmission within 90 days | up to 90 days
  defined as any readmission within 90 days
R0 resection | intraoperative
  defined as tumor-free margins in all the reported surgical margins (biliary and circumferential margins
Intraoperative blood loss | intraoperative
  recorded by the anesthetist using a vacuum system